CLINICAL TRIAL: NCT03277261
Title: Phase III: UbLiTuximab In Multiple Sclerosis Treatment Effects (ULTIMATE I STUDY)
Brief Title: Study to Assess the Efficacy and Safety of Ublituximab in Participants With Relapsing Forms of Multiple Sclerosis (RMS) ( ULTIMATE 1 )
Acronym: ULTIMATE 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TG1101-RMS301; 2017-000638-75 (EudraCT Number)
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Results first posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Relapsing Multiple Sclerosis (RMS)
MeSH Terms: interventions — ublituximab; teriflunomide

STUDY DESIGN:
Intervention Model Description: Randomized, multi-center, double-blinded, active-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded, active-controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ublituximab + Oral Placebo (Experimental): Participants were administered ublituximab 150 milligrams (mg), intravenous (IV) infusion over 4 hours (h) on Day 1 followed by 450 mg over 1 h on Days 15, 168, 336 and 504 (Week 72) along with the oral placebo once daily (QD) from Day 1 up to the last day of Week 95.
  Interventions: Biological: Ublituximab; Drug: Oral Placebo
- Teriflunomide + IV Placebo (Active Comparator): Participants were administered teriflunomide 14 mg tablet, orally, QD from Day 1 up to the last day of Week 95 along with the placebo IV infusion on Days 1, 15, 168, 336 and 504 (Week 72).
  Interventions: Drug: Teriflunomide; Drug: IV Placebo

INTERVENTIONS:
Biological: Ublituximab — Administered as an IV infusion.
  Other Names: TG-1101
  Arms: Ublituximab + Oral Placebo
Drug: Teriflunomide — Film-coated tablets administered orally.
  Arms: Teriflunomide + IV Placebo
Drug: Oral Placebo — Administered orally.
  Arms: Ublituximab + Oral Placebo
Drug: IV Placebo — Administered as an IV infusion.
  Arms: Teriflunomide + IV Placebo

SUMMARY:
This study determines the Annualized Relapse Rate (ARR) in participants with RMS after 96 weeks (approximately 2 years) treatment with intravenous (IV) infusion of ublituximab/oral placebo compared to 14 mg oral teriflunomide/IV placebo.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 age
* Diagnosis of RMS (McDonald criteria 2010)
* Active disease
* Expanded disability status scale (EDSS) 0-5.5 (inclusive) at screening

Exclusion Criteria:

* Treatment with prior Anti-cluster of differentiate 20 (CD20) or other B cell directed treatment
* Treatment with the following therapies at any time prior to randomization: alemtuzumab, natalizumab, teriflunomide, leflunomide and stem cell transplantation
* Diagnosed with Primary Progressive MS (PPMS)
* Pregnant or nursing

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 549 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-11-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - TG Therapeutics RMS Investigational Trial Site, Carlsbad, California
  - TG Therapeutics RMS Investigational Trial Site, Long Beach, California
  - TG Therapeutics RMS Investigational Trial Site, Pasadena, California
  - TG Therapeutics RMS Investigational Trial Site, Stanford, California
  - TG Therapeutics RMS Investigational Trial Site, Miami, Florida
  - TG Therapeutics RMS Investigational Trial Site, Northbrook, Illinois
  - TG Therapeutics RMS Investigational Trial Site, Kansas City, Kansas
  - TG Therapeutics RMS Investigational Trial Site, Detroit, Michigan
  - TG Therapeutics RMS Investigational Trial Site, Amherst, New York
  - TG Therapeutics RMS Investigational Trial Site, Westerville, Ohio
  - TG Therapeutics RMS Investigational Trial Site, Franklin, Tennessee
  - TG Therapeutics RMS Investigational Trial Site, Knoxville, Tennessee
  - TG Therapeutics RMS Investigational Trial Site, Dallas, Texas
  - TG Therapeutics RMS Investigational Site, Round Rock, Texas

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared after study completion via publication.

REFERENCES:
- [Derived] Alvarez E, Steinman L, Fox EJ, Hartung HP, Qian P, Wray S, Robertson D, Selmaj K, Wynn D, Mok K, Xu Y, Bodhinathan K, Miskin HP, Cree BAC. Improvements in no evidence of disease activity with ublituximab vs. teriflunomide in the ULTIMATE phase 3 studies in relapsing multiple sclerosis. Front Neurol. 2024 Oct 24;15:1473284. doi: 10.3389/fneur.2024.1473284. eCollection 2024. PMID 39512280
- [Derived] Steinman L, Fox E, Hartung HP, Alvarez E, Qian P, Wray S, Robertson D, Huang D, Selmaj K, Wynn D, Cutter G, Mok K, Hsu Y, Xu Y, Weiss MS, Bosco JA, Power SA, Lee L, Miskin HP, Cree BAC; ULTIMATE I and ULTIMATE II Investigators. Ublituximab versus Teriflunomide in Relapsing Multiple Sclerosis. N Engl J Med. 2022 Aug 25;387(8):704-714. doi: 10.1056/NEJMoa2201904. PMID 36001711

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 549 participants were enrolled across investigative sites in Belarus, Spain, the United Kingdom, Georgia, Poland, Russia, Serbia, Ukraine, and the United States from 19 September 2017 to 6 November 2020.
Pre-assignment Details: A total of 646 participants were screened and of those, 549 were enrolled and randomized to receive either ublituximab/oral placebo or teriflunomide/IV placebo.
Period: Overall Study
Arm/Group | Ublituximab + Oral Placebo | Teriflunomide + IV Placebo
Started | 274 | 275
Completed (The completed number of participants denote the population who completed the 96 weeks Treatment Period.) | 240 | 252
Not Completed | 34 | 23
Not completed — Adverse Event | 17 | 1
Not completed — Participant Withdrawal of Consent | 6 | 15
Not completed — Investigator / Sponsor Decision | 4 | 2
Not completed — Pregnancy | 2 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Lack of Efficacy | 2 | 2
Not completed — Other-Alternative Treatment/Unspecified Reasons | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat (ITT) population consisted of all randomized participants.
Groups:
- Ublituximab + Oral Placebo: Participants were administered ublituximab 150 mg, IV infusion over 4 h on Day 1 followed by 450 mg over 1 h on Days 15, 168, 336 and 504 (Week 72) along with the oral placebo QD from Day 1 up to the last day of Week 95.
- Total: Total of all reporting groups
Arm/Group | Ublituximab + Oral Placebo | Teriflunomide + IV Placebo | Total
Number analyzed (Participants) | 274 | 275 | 549
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (8.48) | 37.0 (9.62) | 36.7 (9.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167 | 180 | 347
  Male | 107 | 95 | 202
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 2 | 9
  Not Hispanic or Latino | 263 | 267 | 530
  Unknown or Not Reported | 4 | 6 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 6 | 6 | 12
  Race: White | 267 | 267 | 534
  Race: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Race: Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Annualized Relapse Rate (ARR)
Description: ARR is defined as the number of Independent Relapse Adjudication Panel (IRAP)-confirmed relapses per participant year. The estimate of ARR for a treatment group is the total number of relapses for participants in the respective treatment group divided by the sum of treatment duration for participants in that specific treatment group.
Time Frame: Up to 96 weeks
Population: Modified Intention-to-Treat (mITT) population consisted of all participants in the ITT population who received at least one dose of study medication and have at least one baseline and post baseline efficacy assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: relapses per participant-years
Arm/Group | Ublituximab + Oral Placebo | Teriflunomide + IV Placebo
Number analyzed (Participants) | 271 | 274
relapses per participant-years | 0.076 [0.042 to 0.138] | 0.188 [0.124 to 0.283]
Statistical Analysis 1: Comparison: Ublituximab + Oral Placebo vs Teriflunomide + IV Placebo; Test type: Superiority; p < 0.0001, Negative Binomial Model — GEE (Generalized Estimating Equation) model for the relapse count per participant with logarithmic link function, treatment, region, and baseline Expanded Disability Status Scale (EDSS) strata as covariates and log (years of treatment) as offset; Rate Ratio (Ublituximab/Teriflunomide) = 0.406, 95% CI 2-sided [0.268 to 0.615]

2. Secondary Outcome: Total Number of Gadolinium (Gd)-Enhancing T1-Lesions Per Magnetic Resonance Imaging (MRI) Scan Per Participant
Description: The total number of Gd-enhancing T1-lesions were calculated as the sum of the individual number of lesions at Weeks 12, 24, 48, and 96, divided by the total number of MRI scans of the brain.
Time Frame: Weeks 12, 24, 48, and 96
Population: mITT- magnetic resonance imaging (MRI) population included participants in mITT population who have baseline and post-baseline MRI efficacy assessments. Overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: lesions per scan per participant
Arm/Group | Ublituximab + Oral Placebo | Teriflunomide + IV Placebo
Number analyzed (Participants) | 264 | 269
lesions per scan per participant | 0.016 [0.008 to 0.032] | 0.491 [0.355 to 0.679]
Statistical Analysis 1: Comparison: Ublituximab + Oral Placebo vs Teriflunomide + IV Placebo; Test type: Superiority; p < 0.0001, Negative Binomial Model — GEE model for the relapse count per participant with logarithmic link function, treatment, region, and baseline EDSS strata as covariates and log (years of treatment) as offset; Rate Ratio (Ublituximab/Teriflunomide) = 0.033, 95% CI 2-sided [0.019 to 0.058]

3. Secondary Outcome: Total Number of New and Enlarging T2 Hyperintense Lesions (NELs) Per MRI Scan Per Participant
Description: The total number of NELs were calculated as the sum of the individual number of lesions at Weeks 24, 48, and 96, divided by the total number of MRI scans of the brain.
Time Frame: Weeks 24, 48, and 96
Population: mITT- MRI population included participants in mITT population who have baseline and post-baseline MRI efficacy assessments. Overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: lesions per scan per participant
Arm/Group | Ublituximab + Oral Placebo | Teriflunomide + IV Placebo
Number analyzed (Participants) | 260 | 267
lesions per scan per participant | 0.213 [0.144 to 0.316] | 2.789 [2.136 to 3.643]
Statistical Analysis 1: Comparison: Ublituximab + Oral Placebo vs Teriflunomide + IV Placebo; Test type: Superiority; p < 0.0001, Negative Binomial Model — [p-value comment as in outcome 2, analysis 1]; Rate Ratio (Ublituximab/Teriflunomide) = 0.076, 95% CI 2-sided [0.056 to 0.104]

4. Secondary Outcome: Time to Confirmed Disability Progression (CDP) for at Least 12 Weeks
Description: 12-week CDP is defined as an increase in EDSS at least 1 point higher than the baseline EDSS if the baseline EDSS is ≤5.5 or at least 0.5 higher than the baseline EDSS if the baseline EDSS is >5.5. The EDSS is based on a standard neurological examination, (pyramidal, cerebellar, brainstem, sensory, bowel and bladder, visual, and cerebral) and ambulation function system assessments. The EDSS disability scale ranges in 0.5-point steps from 0 (normal) to 10 (death) where higher scores indicate disability. The time to onset of 12-week CDP is the time to progression to the EDSS change defined above.
Time Frame: Up to Week 96
Population: mITT population consisted of all participants in the ITT population who received at least one dose of study medication and have at least one baseline and post baseline efficacy assessment. As per protocol, data was summarized for the mITT Population using pooled data from participants in this study and TG1101-RMS302 [NCT03277248].
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Ublituximab + Oral Placebo | Teriflunomide + IV Placebo
Number analyzed (Participants) | 543 | 546
weeks | NA [NA to NA] — Median and Inter Quartile Range was not reached due to the low number of participants with events. | NA [NA to NA] — Median and Inter Quartile Range was not reached due to the low number of participants with events.

5. Secondary Outcome: Percentage of Participants With No Evidence of Disease Activity (NEDA)
Description: A participant with NEDA is defined as a participant without relapses confirmed by the IRAP, without MRI activities (no T1 Gd+ lesions and no new/enlarging T2 lesions), and no 12-week CDP. Any evidence of disease activity from Week 24 to Week 96 was counted as not reaching NEDA. Any evidence of disease activity before Week 24 was not counted.
Time Frame: Week 24 up to Week 96
Population: mITT population consisted of all participants in the ITT population who received at least one dose of study medication and have at least one baseline and post baseline efficacy assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Ublituximab + Oral Placebo | Teriflunomide + IV Placebo
Number analyzed (Participants) | 271 | 274
percentage of participants | 44.6 | 15.0
Statistical Analysis 1: Comparison: Ublituximab + Oral Placebo vs Teriflunomide + IV Placebo; Test type: Superiority; p < 0.0001, Regression, Logistic — Logistic regression model with treatment, region, baseline EDSS strata and log transformed baseline MRI lesion counts (T1 unenhancing, T2, Gd enhancing) as covariates; Odds Ratio (Ublituximab/Teriflunomide) = 5.442, 95% CI 2-sided [3.536 to 8.375]

6. Secondary Outcome: Percentage of Participants With Impaired Symbol Digit Modalities Test (SDMT)
Description: The SDMT involves a simple substitution task using a reference key, the examinee has 90 seconds to pair specific numbers with given geometric figures. Responses are done verbally. The administration time is approximately 5 minutes. The total SDMT score for each visit ranging from 0-110 is defined as the total number of correct answers reported in the case report form (CRF), where high scores indicate better outcome. Impaired SDMT is defined as a decrease from baseline of at least 4 points at any post-baseline assessment up to the Week 96 visit.
Time Frame: Baseline up to Week 96
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Ublituximab + Oral Placebo | Teriflunomide + IV Placebo
Number analyzed (Participants) | 271 | 274
percentage of participants | 29.2 | 31.8
Statistical Analysis 1: Comparison: Ublituximab + Oral Placebo vs Teriflunomide + IV Placebo; Test type: Superiority; p = 0.4669, Logistic Regression — Logistic regression model with treatment, region, baseline EDSS strata, and log-transformed baseline MRI counts (T1 unenhancing, T2, Gd enhancing) as covariates; Odds Ratio (Ublituximab/Teriflunomide) = 0.872, 95% CI 2-sided [0.603 to 1.261]

7. Secondary Outcome: Percent Change From Baseline in Brain Volume
Time Frame: Baseline up to Week 96
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Ublituximab + Oral Placebo | Teriflunomide + IV Placebo
Number analyzed (Participants) | 204 | 207
percent change | -0.197 [-0.228 to -0.166] | -0.125 [-0.155 to -0.095]
Statistical Analysis 1: Comparison: Ublituximab + Oral Placebo vs Teriflunomide + IV Placebo; Test type: Superiority; p < 0.0001, Mixed Model Repeated Measures (MMRM) — The model includes treatment, region, baseline EDSS strata, visit, treatment-by-visit interaction, and baseline volume (cube root transformed) as covariates and an unstructured covariance matrix; Least squares mean difference = -0.072, 95% CI 2-sided [-0.107 to -0.036]

8. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product. A Serious AE is defined as any untoward medical occurrence that: results in death, is immediately life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, and/or causes a congenital anomaly/birth defect. A TEAE is an AE that starts or worsens after receiving study drug.
Time Frame: From the first dose of study drug through the end of the study (up to approximately 116 weeks)
Population: Safety population included all participants who received at least one dose of study drug (ublituximab or teriflunomide, with corresponding placebos).
Measure: Number; unit: percentage of participants
Arm/Group | Ublituximab + Oral Placebo | Teriflunomide + IV Placebo
Number analyzed (Participants) | 273 | 275
percentage of participants
  TEAEs | 86.1 | 89.1
  TESAEs | 11.4 | 6.9

ADVERSE EVENTS:
Time Frame: From the first dose of study drug through the end of the study (up to approximately 116 weeks)
Description: All-Cause Mortality: All the enrolled participants; Adverse Events: Safety population included all participants who received at least one dose of study drug (ublituximab or teriflunomide, with corresponding placebos).
Arm/Group | Ublituximab + Oral Placebo | Teriflunomide + IV Placebo
All-Cause Mortality (participants affected / at risk) | 2/274 | 0/275
Serious Adverse Events (participants affected / at risk) | 31/273 | 19/275
Other Adverse Events (participants affected / at risk) | 197/273 | 181/275
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ublituximab + Oral Placebo (N=273) | Teriflunomide + IV Placebo (N=275)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 0
COVID-19 pneumonia (Infections and infestations) | 2 | 1
Central nervous system enteroviral infection (Infections and infestations) | 2 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bullous erysipelas (Infections and infestations) | 1 | 0
Encephalitis (Infections and infestations) | 1 | 0
Measles (Infections and infestations) | 1 | 0
Meningoencephalitis viral (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Salpingitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1
Lyme disease (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Neurological symptom (Nervous system disorders) | 1 | 4
Presyncope (Nervous system disorders) | 1 | 0
Acoustic neuritis (Nervous system disorders) | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Affective disorder (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1
Medical device removal (Surgical and medical procedures) | 1 | 0
Varicose vein (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ublituximab + Oral Placebo (N=273) | Teriflunomide + IV Placebo (N=275)
Lymphopenia (Blood and lymphatic system disorders) | 27 | 4
Neutropenia (Blood and lymphatic system disorders) | 11 | 15
Nausea (Gastrointestinal disorders) | 29 | 15
Diarrhoea (Gastrointestinal disorders) | 19 | 26
Abdominal pain upper (Gastrointestinal disorders) | 7 | 14
Pyrexia (General disorders) | 41 | 13
Chills (General disorders) | 19 | 1
Nasopharyngitis (Infections and infestations) | 34 | 44
Respiratory tract infection viral (Infections and infestations) | 20 | 8
Rhinitis (Infections and infestations) | 18 | 8
Urinary tract infection (Infections and infestations) | 11 | 16
Upper respiratory tract infection (Infections and infestations) | 16 | 15
Lymphocyte count decreased (Investigations) | 33 | 8
Aspartate aminotransferase increased (Investigations) | 14 | 4
Alanine aminotransferase increased (Investigations) | 12 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 30
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 12
Headache (Nervous system disorders) | 84 | 59
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 36
Hypertension (Vascular disorders) | 12 | 23
Abdominal pain (Gastrointestinal disorders) | 15 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/61/NCT03277261/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/61/NCT03277261/SAP_001.pdf